CLINICAL TRIAL: NCT00751205
Title: (REASON) Double-blind, Randomized Phase II Study to Evaluate the Safety and Efficacy of Acetyl-l-carnitine in the Prevention of Sagopilone-induced Peripheral Neuropathy.
Brief Title: Prevention of Sagopilone-induced Neurotoxicity With Acetyl-L-Carnitine (ALC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91695; 2008-000879-26 (EudraCT Number)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer; Ovarian Cancer
Keywords: Peripheral Neuropathy; Prostate Carcinoma; Ovarian Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Ovarian Neoplasms; Peripheral Nervous System Diseases | interventions — sagopilone; Acetylcarnitine; allantoicase; Prednisolone; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sagopilone 16 mg/m^2 i.v., Acetyl-L-Carnitine (ALC) 1000 mg tid, HRPC only: Prednisone or Prednisolone 5 mg bid
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Sagopilone 16 mg/m^2 i.v. and placebo 1000 mg tid, HRPC only: Prednisone or Prednisolone 5 mg bid

INTERVENTIONS:
Drug: Sagopilone 16 mg/m^2 i.v., Acetyl-L-Carnitine (ALC) 1000 mg tid, HRPC only: Prednisone or Prednisolone 5 mg bid — Subjects will receive intravenous (i.v.) infusion of Sagopilone for 3 hours on day 1 of a 3-weeks cycle. In addition, subjects will receive Acetyl-L-Carnitine (ALC) 1000 mg tid. Treatment with Sagopilone and ALC will be continued as long as there is benefit. Subjects with HRPC will also receive Prednisone or Prednisolone 5 mg bid, throughout the treatment with Sagopilone.
  Arms: Arm 1
Drug: Sagopilone 16 mg/m^2 i.v. and placebo 1000 mg tid, HRPC only: Prednisone or Prednisolone 5 mg bid — Subjects will receive intravenous (i.v.) infusion of Sagopilone for 3 hours on day 1 of a 3-weeks cycle. Treatment will be continued as long as there is benefit. In addition, subjects will receive 21 weeks of placebo 1000 mg tid. After all patients have completed 6 cycles of treatment, an analysis will be performed to see whether ALC was better than placebo. If this is the case, patients still under placebo treatment will be offered to switch to ALC. Subjects with HRPC will also receive Prednisone or Prednisolone 5 mg bid, throughout the treatment with Sagopilone.
  Arms: Arm 2

SUMMARY:
This study investigates the safety and efficacy of Acetyl-L-Carnitine and compares it to the safety and efficacy of a placebo (inactive) tablet in the prevention of Sagopilone-induced peripheral neuropathy. Patients will receive intravenous infusion of sagopilone for 3 hours on day 1 of a 3-weeks cycle. Treatment with Sagopilone will be given as long as the patient is benefitting. In addition patients will receive ALC or placebo, starting 1 week before first sagopilone infusion and ending 30-33 days after the last infusion with sagopilone. Safety will be determined by laboratory and other evaluations. Efficacy of ALC will be determined by the incidence of all grades of peripheral neuropathy with the results of a patient questionnaire. Efficacy of the combination of ALC and Sagopilone will be determined by the tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged >/= 18 years
* Epithelial ovarian, peritoneal cavity or Fallopian tube cancer (except mucinous or clear cell tumors) or Adenocarcinoma of the prostate
* At least 1 unidimensional measurable lesion (suitable for RECIST evaluation) or for patients without measurable disease, CA 125 levels >/= 2 times the upper limit of normal (ULN) within 3 months and confirmed within 2 weeks prior to first infusion (ovarian cancer) or PSA value >/= 5 ng/mL (HRPC).
* Progression of disease (HRPC) despite adequate androgen-inhibiting hormone therapy.
* Progression of disease (Ovarian Cancer) or symptomatic relapse after previous therapy (elevated CA125 levels alone are insufficient for inclusion) WHO performance status 0 to 1
* No clinical residual neuropathy (CTCAE Grade 0 at baseline)
* Adequate recovery from previous surgery, radiation, and chemotherapy (excluding alopecia)
* Adequate function of major organs and systems.
* Survival expectation =3 months
* Histologically or cytologically proven:

  1. Epithelial ovarian, peritoneal cavity or Fallopian tube cancer (except mucionous cell tumors or clear cell tumors that have a clear cell component of >33%)

Exclusion Criteria:

* Symptomatic brain metastases requiring whole- brain irradiation
* Any concomitant malignancy: the following exceptions are allowed: Non-melanoma skin cancer, Carcinoma in situ of the cervix, Malignancy with definitive treatment >/= 5 years ago without relapse.
* Diabetes mellitus (even if controlled only by special diet)
* History of chronic hepatitis B or C, or known HIV infection
* Seizure disorder requiring medication (such as steroids or anti-epileptics)
* Inability to swallow oral medications
* Prior treatment with epothilones
* Concomitant use of neurotoxic drugs
* Concomitant use of compounds that have potentially positive effects towards symptoms of neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Overall incidence of peripheral neuropathy (any grade) during at most 6 cycles of Sagopilone treatment, based on the Adverse Events. | Start of Sagopilone treatment until at most 6 cycles + 1 month.

SECONDARY OUTCOMES:
Efficacy of ALC: incidence of neuropathy of grade 3 or 4, time to onset of neuropathy, duration of neuropathy. | Start of treatment to safety Follow-up
Efficacy of ALC: Percentage of discontinuations due to neuropathy. | Start of treatment to safety Follow-up
Safety of Sagopilone in combination with ALC. | Baseline to Safety follow-up
Efficacy of Sagopilone: 'best overall response' according to modRECIST criteria | Start treatment to End of Treatment
Efficacy of Sagopilone: 'best overall response' according to CA-125 or PSA response | Start treatment to End of Treatment
Efficacy of Sagopilone: Time to disease progression, Progression-free survival | Start treatment to Progression or Death
Efficacy of Sagopilone: Duration of response | Start treatment to Progression or Death
Efficacy of Sagopilone: WHO performance status. | Screening to end of Treatment
Pharmacokinetic: Sagopilone concentrations (optional) | Day 1,2,3,5,15 of cycle 1 and day2
Pharmacokinetic: ALC concentrations | radomisation, day 1 of cycle 1 and 2
Pharmacogenomics (optional): in tumor tissue, blood and ascites | Blood sample at screening, tissue sample and ascites whenever available

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Bruxelles - Brussel, Belgium
- France (5):
  - Caen
  - Montpellier
  - Nantes
  - Paris
  - Villejuif
- Germany (5):
  - Tübingen, Baden-Wurttemberg
  - Rostock, Mecklenburg-Vorpommern
  - Bonn, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Magdeburg, Saxony-Anhalt
- Italy (4):
  - Meldola, Forlì
  - Bologna
  - Rimini
  - Roma
- Netherlands (3):
  - Amsterdam
  - Leiden
  - Maastricht
- United Kingdom (2):
  - Leicester, Leicestershire
  - Northwood, Middlesex

REFERENCES:
- [Derived] Campone M, Berton-Rigaud D, Joly-Lobbedez F, Baurain JF, Rolland F, Stenzl A, Fabbro M, van Dijk M, Pinkert J, Schmelter T, de Bont N, Pautier P. A double-blind, randomized phase II study to evaluate the safety and efficacy of acetyl-L-carnitine in the prevention of sagopilone-induced peripheral neuropathy. Oncologist. 2013;18(11):1190-1. doi: 10.1634/theoncologist.2013-0061. Epub 2013 Oct 8. PMID 24105751
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/